CLINICAL TRIAL: NCT04876339
Title: Sonification Techniques for Gait Training: a Pilot Multicentric Randomized Controlled Trial
Brief Title: Sonification Techniques for Gait Training
Acronym: SonicWalk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2419 CE
Record Dates: First submitted 2021-04-26; First posted 2021-05-06 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease; Stroke; Multiple Sclerosis
MeSH Terms: conditions — Parkinson Disease; Stroke; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gait rehabilitation with "sonification" (Experimental): The rehabilitation exercises with sonification are supported by the musical component (see "Interventions" section for details).
  Interventions: Device: Gait rehabilitation with "sonification"
- Standard gait rehabilitation (without sonification) (Active Comparator): The same rehabilitation exercises are performed without musical support.
  Interventions: Other: Standard gait rehabilitation (without sonification)

INTERVENTIONS:
Device: Gait rehabilitation with "sonification" — The sonification system is composed by 2 inertial sensors, a computer and a pair of bluetooth headphones connected with the computer. The sensors will be placed one per leg at the ankle and connected with Matlab software. An home-made ad-hoc software associates patient's movements with music patterns. The patient's natural rhythm is detected and used at the beginning of the intervention. The first part of each exercise is supported by a pre-recorded chord progression with a click on the background. In the second part (sonification approach) the software notices and records the contact of the heel with the ground. Each contact activates musical stimuli listened to via headphones. The steps succession will build a regular and predictable musical progression in relation to the correct sequence of steps. The exercises planned in this intervention are the same as those planned in the gait standard rehabilitation (see below).
  Arms: Gait rehabilitation with "sonification"
Other: Standard gait rehabilitation (without sonification) — The training will be carried out without any musical support. Exercises I Phase
  1. Load shift in anteroposterior standing in tandem position, left foot forward (3 minutes exercise with a short break in the middle)
  2. Load shift in anteroposterior standing in tandem position, right foot forward (3 minutes exercise with a short break in the middle)
  3. Left foot swing (3 minutes exercise with a short break in the middle)
  4. Right foot swing (3 minutes exercise with a short break in the middle)
  5. March in place (3 minutes exercise with a short break in the middle) Exercises II phase (15 minutes): the patient will perform 14 minutes of walking with a 1 minute of break in the middle (7 minutes of walking, 1 minute rest, 7 minutes of walking). In the second part of walking the patient will be asked to slightly increase the pace of the step up to the maximum possible speed.
  Arms: Standard gait rehabilitation (without sonification)

SUMMARY:
Music therapy is widely used in relational and rehabilitation settings. In addition to Neurologic Music Therapy and other music-based techniques, "sonification" approaches were recently introduced in the field of rehabilitation. The "sonification" can be defined as a properly selected set of sonorous-music stimuli are associated with patient movements mapping. In fact, the auditory-motor feedback can replace damaged proprioceptive circuits with a consequent improvement of the rehabilitation process. Interventions with "sonification" facilitate sensorimotor learning, proprioception and movements planning and execution improving global motor parameters. This study proposes the use of musical auditory cues which includes the melodic-harmonic component of the music. This kind of sonification makes the feedback pleasant and predictable as well as potentially effective. The investigators propose to apply and assess the effectiveness of this kind of sonification on gait training and other secondary outcomes in stroke, Parkinson's disease and multiple sclerosis population. Also, the investigators will assess the impact of "sonification" on the level of fatigue perceived during the rehabilitation process and on the quality of life. The study is a multicenter randomized controlled trial and will involve 120 patients that will undergo standard motor rehabilitation or the same rehabilitation but with the sonification support. The interventions will be evaluated at the baseline, after 10 sessions, after 20 sessions and at follow-up (one month after the end of the treatment). The assessment will include functional, motor, fatigue and quality of life evaluations. The collected data will be statistically processed.

DETAILED DESCRIPTION:
Background:

Music therapy is widely used in relational settings. The sound can engage limbic and paralimbic areas and a variety of other brain areas strictly connected with movement (motor cortex, supplementary motor area, cerebellum, basal ganglia, etc.). For this reason, music can be considered a useful tool in rehabilitation settings and, in particular, for neuromotor rehabilitation.

The use of specific music-based techniques can induce plastic changes from childhood to elderly. These changes involve both brain motor and auditory sensory-motor areas thanks to the improved connectivity between brain areas induced by the sound and music that would not happen without the auditory stimuli. As suggested in previous studies the plastic changes induced by music in the nodal points of the cerebral network can cause effects that tend to persist even beyond the duration of rehabilitation training. The music also in the rehabilitation process determines an emotional involvement and creates a strong motivational basis reinforcing its action through the coupling of the auditory stimulus with sensory-motor component.

Neurologic Music Therapy (NTM) could be defined as a codified use of music-based techniques aimed at recovering sensory, cognitive and motor deficits due to a neurological pathology. NMT consists in several specific techniques among which Rhythmic Auditory Stimulation (RAS) is one of the most used and well documented in scientific literature. RAS is based on the application of the rhythmic component of the music to gait and gait-related rehabilitation. Music effects in stroke rehabilitation are well documented: music can improve gait (velocity, cadence, stride length and balance), upper limbs movements , language, but also mood and psychological aspects.

Gait rehabilitation studies for Parkinson's Disease (PD) and Multiple Sclerosis (MS) show similar results.

Recent studies are related to the "sonification" technique: a properly selected set of sonorous-music stimuli are associated with patient movements mapping. The auditory-motor feedback can replace damaged proprioceptive circuits with a consequent improvement of the rehabilitation process. Interventions with "sonification" facilitate sensorimotor learning, proprioception and movements planning and execution improving global motor parameters. Studies related to "sonification" mainly concern upper limb rehabilitation and only a few of them concern the lower limbs rehabilitation. In particular, this study proposes the use of musical auditory cues which includes the melodic-harmonic component of the music. This kind of sonification makes the feedback pleasant and predictable as well as potentially effective. The investigators propose to apply this particular kind of sonification to gait training and other secondary outcomes in stroke, PD and SM population.

Aims:

1. To assess the effectiveness of the sonification in the gait rehabilitation in stroke, PD and MS patients.
2. To assess the effectiveness of sonification on the level of fatigue perceived during the rehabilitation process
3. To assess the impact of the sonification on the quality of life

Materials and methods:

The study is a multicenter randomized controlled trial and will involve 120 clinically stabilized patients with stroke (n=40), Parkinsons' disease (n=40) and multiple sclerosis (n=40). Each of these three arms will be divided in two groups: a control group (n=20) will undergo standard motor rehabilitation and an experimental group (n=20) will undergo the same rehabilitation but with the sonification support. The gait training program includes 20 sessions, 30 minutes each 3 times a week (see next chapter for details).

A unique randomization list will be generated according to the trial's design and managed by the Principal Investigator. Each subject will be associated with a unique identifier that will allow its identification throughout the duration of the study. The evaluation of the questionnaires and the statistical analysis will be carried out blindly

Assessment:

The interventions will be evaluated at the baseline (T0), after 10 sessions (T1), after 20 sessions (T2, end of the treatment) and at follow-up (T3, one month after the end of the treatment). The scales used for the assessments will be the following:

Functional evaluation:

- Functional Independence Measure (FIM)

Motor parameter evaluation:

* 6 minutes Walking Test (velocity)
* Mini BesTest (balance)
* Dynamic Gait Index (dynamic balance, gait and risk of falls)
* Timed Up & Go (mobility)

Fatigue assessments, quality of life and perceived overall effect of the intervention:

* VAS (Visual Analogue Scale, for assessing perceived fatigue at the end of each session)
* McGill Quality of Life- it (quality of life assessment)
* Global Perceived Effect (GPE) Statistics The collected data will be presented by descriptive statistics: continuous variables having a normal distribution as mean and standard deviation, continuous variables having a non-normal distribution as median and interquartile range. Binary and categorical variables will be presented as a percentage or absolute number.

For each group of patients involved in this study (stroke, Parkinson's disease, multiple sclerosis), the homogeneity of demographic data and outcome measures between the experimental subgroup and the control subgroup will be verified. Finally, for all outcome measures detected (6 minutes Walking Test, FIM, Dynamic Gait Index, Timed Up & Go, VAS fatigue, McGill Quality of Life-it and GPE) it is expected to perform the analysis of the variance or mixed linear model for repeated measurements (p<0.05) in order to evaluate the effects of the treatment type, time and their interaction. For those outcomes where the assumptions of applicability of the variance analysis will not be verified, non-parametric methods will be applied to assess the main effects and interaction separately.

Patients will be asked to sign an Informed Consent before joining the study.

Adverse events No indication of any risk associated with the protocol because the rehabilitative treatments will be performed according to the usual procedures laid down in clinical practice in accordance with the guidelines relating to the gait rehabilitation.

Informed consent to participate in the study. All patients participating in the study will have to give their informed consent as required by the attachment for the execution of the study and for the processing of personal data.

Insurance The activation of an additional insurance is not foreseen as the study and the procedures applied fall within the coverage of the insurance policy currently in force for the conduct of the clinical trial.

ELIGIBILITY:
Inclusion criteria (stroke patients)

* Age < 80
* Mini Mental State Examination > 24
* Modified Rankin Scale: 1-3
* Single hemisphere lesion
* Stabilized disease (> 6 months after the acute event)
* Impairment in gait parameters (e.g. velocity, perceived fatigue etc)
* Motor independence during walking (without orthotic devices and aids) but with pathological pattern (spasticity level: Ashworth < 2)

Inclusion criteria (patients with Parkinson's disease)

* Age < 80
* Mini Mental State Examination > 24
* Unified Parkinson Disease Rating Scale score (Parte III): < 28
* Stabilized disease and drug therapy
* Altered gait patterns
* Motor independence during walking (without orthotic devices and aids) but with pathological pattern

Inclusion criteria (patients with multiple sclerosis):

* Age < 60
* Mini Mental State Examination > 24
* Expanded Disability Status Scale score: 3-5
* Stabilized disease in the last 6 months (without relapse or disability progression)
* Altered gait patterns (i.e., careening, slowing down, spasticity: Ashworth < 2, etc.)
* Motor independence during walking

Exclusion Criteria (stroke patients)

* Multiple or bilateral lesions
* Neglect
* Equinism
* Spasticity: Ashworth >2
* Structured (non-elastic) Achilles tendon retraction
* Neurotoxin in the 3 months prior to the study
* Baclofen introduced or modified in the week before the start of the study
* Previous or concurrent diseases disabling the lower limb functions
* Rehabilitative treatments with music in the year before the study

Exclusion criteria (patients with Parkinson's disease):

* Previous or concurrent diseases disabling the lower limb functions
* Changes of drug therapy during the study
* Rehabilitative treatments with music in the year before the study

Exclusion criteria (patients with multiple sclerosis):

* Previous or concurrent diseases disabling the lower limb functions
* Neurotoxin in the 3 months prior to the study
* Baclofen introduced or modified in the week before the start of the study
* Spasticity: Ashworth >2
* Structured (non-elastic) Achilles tendon retraction
* Rehabilitative treatments with music in the year before the study

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Six Minutes Walking Test | Change from Baseline Six Minutes Walking Test at 7 weeks
  The gait speed will be evaluated (using the Six Minutes Walking Test) by comparing the variations of the test scores in the experimental and control group

SECONDARY OUTCOMES:
Mini BesTest | Up to 11 weeks
  The balance will be evaluated (using the Mini BesTest) by comparing the variations of the test scores in the experimental and control group
Dynamic Gait Index | Up to 11 weeks
  Dynamic balance and gait and risk of falls will be evaluated (using the Dynamic Gait Index) by comparing the variations of the test scores in the experimental and control group
Timed Up & Go | Up to 11 weeks
  The mobility will be evaluated (using the Timed Up & Go test) by comparing the variations of the test scores in the experimental and control group

OTHER OUTCOMES:
McGill Quality of Life- it | Up to 11 weeks
  Quality of Life will be evaluated (using the McGill Quality of Life- it) by comparing the variations of the test scores in the experimental and control group
Global Perceived Effect | Up to 11 weeks
  The overall effect of the intervention will be evaluated (using the Global Perceived Effect) by comparing the variations of the test scores in the experimental and control group
Visual Analogue Scale | Up to 11 weeks
  The fatigue perceived will be evaluated (using a Visual Analogue Scale) by comparing the variations of the test scores in the experimental and control group

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Raglio, PhD, Principal Investigator — Istituti Clinici Scientifici Maugeri IRCCS, Pavia, Italy
Locations (1):
- Istituti Clinici Scientifici Maugeri IRCCS, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altenmuller E, Marco-Pallares J, Munte TF, Schneider S. Neural reorganization underlies improvement in stroke-induced motor dysfunction by music-supported therapy. Ann N Y Acad Sci. 2009 Jul;1169:395-405. doi: 10.1111/j.1749-6632.2009.04580.x. PMID 19673814
- [Background] Ashoori A, Eagleman DM, Jankovic J. Effects of Auditory Rhythm and Music on Gait Disturbances in Parkinson's Disease. Front Neurol. 2015 Nov 11;6:234. doi: 10.3389/fneur.2015.00234. eCollection 2015. PMID 26617566
- [Background] Bangert M, Altenmuller EO. Mapping perception to action in piano practice: a longitudinal DC-EEG study. BMC Neurosci. 2003 Oct 15;4:26. doi: 10.1186/1471-2202-4-26. PMID 14575529
- [Background] Bangert M, Peschel T, Schlaug G, Rotte M, Drescher D, Hinrichs H, Heinze HJ, Altenmuller E. Shared networks for auditory and motor processing in professional pianists: evidence from fMRI conjunction. Neuroimage. 2006 Apr 15;30(3):917-26. doi: 10.1016/j.neuroimage.2005.10.044. Epub 2005 Dec 27. PMID 16380270
- [Background] Baram Y, Miller A. Auditory feedback control for improvement of gait in patients with Multiple Sclerosis. J Neurol Sci. 2007 Mar 15;254(1-2):90-4. doi: 10.1016/j.jns.2007.01.003. Epub 2007 Feb 20. PMID 17316692
- [Background] Baumann S, Koeneke S, Schmidt CF, Meyer M, Lutz K, Jancke L. A network for audio-motor coordination in skilled pianists and non-musicians. Brain Res. 2007 Aug 3;1161:65-78. doi: 10.1016/j.brainres.2007.05.045. Epub 2007 Jun 4. PMID 17603027
- [Background] Bella SD, Benoit CE, Farrugia N, Keller PE, Obrig H, Mainka S, Kotz SA. Gait improvement via rhythmic stimulation in Parkinson's disease is linked to rhythmic skills. Sci Rep. 2017 Feb 24;7:42005. doi: 10.1038/srep42005. PMID 28233776
- [Background] Bevilacqua F, Boyer EO, Francoise J, Houix O, Susini P, Roby-Brami A, Hanneton S. Sensori-Motor Learning with Movement Sonification: Perspectives from Recent Interdisciplinary Studies. Front Neurosci. 2016 Aug 25;10:385. doi: 10.3389/fnins.2016.00385. eCollection 2016. PMID 27610071
- [Background] Brodie MA, Dean RT, Beijer TR, Canning CG, Smith ST, Menant JC, Lord SR. Symmetry matched auditory cues improve gait steadiness in most people with Parkinson's disease but not in healthy older people. J Parkinsons Dis. 2015;5(1):105-16. doi: 10.3233/JPD-140430. PMID 25468233
- [Background] Cha Y, Kim Y, Hwang S, Chung Y. Intensive gait training with rhythmic auditory stimulation in individuals with chronic hemiparetic stroke: a pilot randomized controlled study. NeuroRehabilitation. 2014;35(4):681-8. doi: 10.3233/NRE-141182. PMID 25318784
- [Background] Chong HJ, Han SJ, Kim YJ, Park HY, Kim SJ. Relationship between output from MIDI-keyboard playing and hand function assessments on affected hand after stroke. NeuroRehabilitation. 2014;35(4):673-80. doi: 10.3233/NRE-141166. PMID 25318775
- [Background] Colombo R, Raglio A, Panigazzi M, Mazzone A, Bazzini G, Imarisio C, Molteni D, Caltagirone C, Imbriani M. The SonicHand Protocol for Rehabilitation of Hand Motor Function: A Validation and Feasibility Study. IEEE Trans Neural Syst Rehabil Eng. 2019 Apr;27(4):664-672. doi: 10.1109/TNSRE.2019.2905076. Epub 2019 Mar 14. PMID 30872238
- [Background] Conklyn D, Stough D, Novak E, Paczak S, Chemali K, Bethoux F. A home-based walking program using rhythmic auditory stimulation improves gait performance in patients with multiple sclerosis: a pilot study. Neurorehabil Neural Repair. 2010 Nov-Dec;24(9):835-42. doi: 10.1177/1545968310372139. Epub 2010 Jul 19. PMID 20643882
- [Background] Ghai S, Ghai I. Effects of (music-based) rhythmic auditory cueing training on gait and posture post-stroke: A systematic review & dose-response meta-analysis. Sci Rep. 2019 Feb 18;9(1):2183. doi: 10.1038/s41598-019-38723-3. PMID 30778101
- [Background] Ghai S, Ghai I, Schmitz G, Effenberg AO. Effect of rhythmic auditory cueing on parkinsonian gait: A systematic review and meta-analysis. Sci Rep. 2018 Jan 11;8(1):506. doi: 10.1038/s41598-017-16232-5. PMID 29323122
- [Background] Hayden R, Clair AA, Johnson G, Otto D. The effect of rhythmic auditory stimulation (RAS) on physical therapy outcomes for patients in gait training following stroke: a feasibility study. Int J Neurosci. 2009;119(12):2183-95. doi: 10.3109/00207450903152609. PMID 19916847
- [Background] Hausdorff JM, Lowenthal J, Herman T, Gruendlinger L, Peretz C, Giladi N. Rhythmic auditory stimulation modulates gait variability in Parkinson's disease. Eur J Neurosci. 2007 Oct;26(8):2369-75. doi: 10.1111/j.1460-9568.2007.05810.x. PMID 17953624
- [Background] Kim SJ, Koh I. The effects of music on pain perception of stroke patients during upper extremity joint exercises. J Music Ther. 2005 Spring;42(1):81-92. doi: 10.1093/jmt/42.1.81. PMID 15839735
- [Background] Kim DS, Park YG, Choi JH, Im SH, Jung KJ, Cha YA, Jung CO, Yoon YH. Effects of music therapy on mood in stroke patients. Yonsei Med J. 2011 Nov;52(6):977-81. doi: 10.3349/ymj.2011.52.6.977. PMID 22028163
- [Background] Kim SJ, Jo U. Study of accent-based music speech protocol development for improving voice problems in stroke patients with mixed dysarthria. NeuroRehabilitation. 2013;32(1):185-90. doi: 10.3233/NRE-130835. PMID 23422471
- [Background] Jun EM, Roh YH, Kim MJ. The effect of music-movement therapy on physical and psychological states of stroke patients. J Clin Nurs. 2013 Jan;22(1-2):22-31. doi: 10.1111/j.1365-2702.2012.04243.x. Epub 2012 Sep 17. PMID 22978325
- [Background] Lim KB, Kim YK, Lee HJ, Yoo J, Hwang JY, Kim JA, Kim SK. The therapeutic effect of neurologic music therapy and speech language therapy in post-stroke aphasic patients. Ann Rehabil Med. 2013 Aug;37(4):556-62. doi: 10.5535/arm.2013.37.4.556. Epub 2013 Aug 26. PMID 24020037
- [Background] Magee WL, Davidson JW. The effect of music therapy on mood states in neurological patients: a pilot study. J Music Ther. 2002 Spring;39(1):20-9. doi: 10.1093/jmt/39.1.20. PMID 12015809
- [Background] Meyer M, Elmer S, Baumann S, Jancke L. Short-term plasticity in the auditory system: differential neural responses to perception and imagery of speech and music. Restor Neurol Neurosci. 2007;25(3-4):411-31. PMID 17943016
- [Background] Moumdjian L, Moens B, Maes PJ, Van Geel F, Ilsbroukx S, Borgers S, Leman M, Feys P. Continuous 12 min walking to music, metronomes and in silence: Auditory-motor coupling and its effects on perceived fatigue, motivation and gait in persons with multiple sclerosis. Mult Scler Relat Disord. 2019 Oct;35:92-99. doi: 10.1016/j.msard.2019.07.014. Epub 2019 Jul 20. PMID 31357124
- [Background] Moumdjian L, Moens B, Maes PJ, Van Nieuwenhoven J, Van Wijmeersch B, Leman M, Feys P. Walking to Music and Metronome at Various Tempi in Persons With Multiple Sclerosis: A Basis for Rehabilitation. Neurorehabil Neural Repair. 2019 Jun;33(6):464-475. doi: 10.1177/1545968319847962. Epub 2019 May 13. PMID 31079541
- [Background] Purdie H, Hamilton S, Baldwin S. Music therapy: facilitating behavioural and psychological change in people with stroke--a pilot study. Int J Rehabil Res. 1997 Sep;20(3):325-7. No abstract available. PMID 9331582
- [Background] Rodger MW, Young WR, Craig CM. Synthesis of walking sounds for alleviating gait disturbances in Parkinson's disease. IEEE Trans Neural Syst Rehabil Eng. 2014 May;22(3):543-8. doi: 10.1109/TNSRE.2013.2285410. Epub 2013 Oct 25. PMID 24235275
- [Background] Sarkamo T, Tervaniemi M, Laitinen S, Forsblom A, Soinila S, Mikkonen M, Autti T, Silvennoinen HM, Erkkila J, Laine M, Peretz I, Hietanen M. Music listening enhances cognitive recovery and mood after middle cerebral artery stroke. Brain. 2008 Mar;131(Pt 3):866-76. doi: 10.1093/brain/awn013. PMID 18287122
- [Background] Sarkamo T, Pihko E, Laitinen S, Forsblom A, Soinila S, Mikkonen M, Autti T, Silvennoinen HM, Erkkila J, Laine M, Peretz I, Hietanen M, Tervaniemi M. Music and speech listening enhance the recovery of early sensory processing after stroke. J Cogn Neurosci. 2010 Dec;22(12):2716-27. doi: 10.1162/jocn.2009.21376. PMID 19925203
- [Background] Schlaug G. Part VI introduction: listening to and making music facilitates brain recovery processes. Ann N Y Acad Sci. 2009 Jul;1169:372-3. doi: 10.1111/j.1749-6632.2009.04869.x. No abstract available. PMID 19673811
- [Background] Schneider S, Schonle PW, Altenmuller E, Munte TF. Using musical instruments to improve motor skill recovery following a stroke. J Neurol. 2007 Oct;254(10):1339-46. doi: 10.1007/s00415-006-0523-2. Epub 2007 Jan 27. PMID 17260171
- [Background] Scholz DS, Rohde S, Nikmaram N, Bruckner HP, Grossbach M, Rollnik JD, Altenmuller EO. Sonification of Arm Movements in Stroke Rehabilitation - A Novel Approach in Neurologic Music Therapy. Front Neurol. 2016 Jun 30;7:106. doi: 10.3389/fneur.2016.00106. eCollection 2016. PMID 27445970
- [Background] Scholz DS, Rhode S, Grossbach M, Rollnik J, Altenmuller E. Moving with music for stroke rehabilitation: a sonification feasibility study. Ann N Y Acad Sci. 2015 Mar;1337:69-76. doi: 10.1111/nyas.12691. PMID 25773619
- [Background] Scholz DS, Wu L, Pirzer J, Schneider J, Rollnik JD, Grossbach M, Altenmuller EO. Sonification as a possible stroke rehabilitation strategy. Front Neurosci. 2014 Oct 20;8:332. doi: 10.3389/fnins.2014.00332. eCollection 2014. PMID 25368548
- [Background] Shahraki M, Sohrabi M, Taheri Torbati HR, Nikkhah K, NaeimiKia M. Effect of rhythmic auditory stimulation on gait kinematic parameters of patients with multiple sclerosis. J Med Life. 2017 Jan-Mar;10(1):33-37. PMID 28255373
- [Background] Suh JH, Han SJ, Jeon SY, Kim HJ, Lee JE, Yoon TS, Chong HJ. Effect of rhythmic auditory stimulation on gait and balance in hemiplegic stroke patients. NeuroRehabilitation. 2014;34(1):193-9. doi: 10.3233/NRE-131008. PMID 24284453
- [Background] Tamplin J, Baker FA, Jones B, Way A, Lee S. 'Stroke a Chord': the effect of singing in a community choir on mood and social engagement for people living with aphasia following a stroke. NeuroRehabilitation. 2013;32(4):929-41. doi: 10.3233/NRE-130916. PMID 23867418
- [Background] Thaut MH, McIntosh GC, Rice RR. Rhythmic facilitation of gait training in hemiparetic stroke rehabilitation. J Neurol Sci. 1997 Oct 22;151(2):207-12. doi: 10.1016/s0022-510x(97)00146-9. PMID 9349677
- [Background] Thaut MH. Rhythm, music and the brain: Scientific foundations and Clinical applications. New York and London: Taylor & Francis Group; 2005.
- [Background] Thaut MH, Leins AK, Rice RR, Argstatter H, Kenyon GP, McIntosh GC, Bolay HV, Fetter M. Rhythmic auditory stimulation improves gait more than NDT/Bobath training in near-ambulatory patients early poststroke: a single-blind, randomized trial. Neurorehabil Neural Repair. 2007 Sep-Oct;21(5):455-9. doi: 10.1177/1545968307300523. Epub 2007 Apr 10. PMID 17426347
- [Background] van Delden AL, Peper CL, Nienhuys KN, Zijp NI, Beek PJ, Kwakkel G. Unilateral versus bilateral upper limb training after stroke: the Upper Limb Training After Stroke clinical trial. Stroke. 2013 Sep;44(9):2613-6. doi: 10.1161/STROKEAHA.113.001969. Epub 2013 Jul 18. PMID 23868279
- [Background] van Wijck F, Knox D, Dodds C, Cassidy G, Alexander G, MacDonald R. Making music after stroke: using musical activities to enhance arm function. Ann N Y Acad Sci. 2012 Apr;1252:305-11. doi: 10.1111/j.1749-6632.2011.06403.x. PMID 22524372
- [Background] Villeneuve M, Penhune V, Lamontagne A. A piano training program to improve manual dexterity and upper extremity function in chronic stroke survivors. Front Hum Neurosci. 2014 Aug 22;8:662. doi: 10.3389/fnhum.2014.00662. eCollection 2014. PMID 25202258
- [Background] Wolpert DM, Ghahramani Z. Computational principles of movement neuroscience. Nat Neurosci. 2000 Nov;3 Suppl:1212-7. doi: 10.1038/81497. PMID 11127840
- [Background] Wittwer JE, Webster KE, Hill K. Rhythmic auditory cueing to improve walking in patients with neurological conditions other than Parkinson's disease--what is the evidence? Disabil Rehabil. 2013 Jan;35(2):164-76. doi: 10.3109/09638288.2012.690495. Epub 2012 Jun 8. PMID 22681598